CLINICAL TRIAL: NCT02204631
Title: A Two-phase Study to Evaluate the Use of Educational Materials in the Head and Neck Cancer Center
Brief Title: 2 Phase Use Of Educational Materials In Head And Neck Cancer Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-244
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Head and Neck Educational Handbook (Experimental): * Prior to starting treatment, patients will be approached for trial participation and baseline questionnaires (demographics, psychological distress, symptom burden, and illness perception).
  * After enrollment and baseline data collection, the participant will be given the handbook. The clinician giving out the handbook will give an overview of the handbook and flip through the important sections. The clinician will encourage the participant to bring it back and forth.
  * Participants will complete questionnaires at 3 weeks into treatment and 2 weeks after treatment has ended (information satisfaction, psychological distress, symptom burden, and illness perception).
  Interventions: Other: Head and Neck Educational Handbook
- Non Head and Neck Educational Handbook (No Intervention): * Prior to starting treatment, patients will be approached for trial participation and baseline questionnaires (demographics, psychological distress, symptom burden, and illness perception).
  * The first group of participants will not receive the handbook but will receive the current standard care in the head and neck disease center.
  * Participants will complete questionnaires at 3 weeks into treatment and 2 weeks after treatment has ended (information satisfaction, psychological distress, symptom burden, and illness perception).
  * At completion of "Phase I", all 30 participants will also be given a copy of the handbook and an accompanying questionnaire.

INTERVENTIONS:
Other: Head and Neck Educational Handbook
  Arms: Head and Neck Educational Handbook

SUMMARY:
The goal of this study is to assess the experience of our patients with head and neck cancer in regard to the information they receive, their symptoms, and their understanding of their diagnosis, to determine ways to improve upon these aspects of patient care in the future.

DETAILED DESCRIPTION:
There will be two phases of the study. In "Phase I", 30 participants will be recruited for assessment of information satisfaction, psychological stress, illness perception, and symptom burden throughout their head and neck cancer treatment without any intervention. This group will represent the current standard of care in the head and neck group and serve as a "historical control" for the second group. In "Phase II", which will occur after "Phase I" group, 30 new participants will be recruited to receive a handbook and to have it integrated into their cancer care. The same participant reported outcome measures of information satisfaction, psychological stress, illness perception, and symptom burden will be assessed such that comparisons between phases can be made. This will serve as a pilot study of the implementation and maintenance of an educational intervention in clinical practice and how it affects participant-reported outcomes. Comparison of these two groups of participants will provide the baseline data to plan future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years old) with a new diagnosis of head and neck cancer.
* Patients who have a treatment plan including both chemotherapy and radiation.
* Patients who will be undergoing treatment at Massachusetts General Hospital Cancer Center.
* Ability to speak and read in English in order to be able to complete questionnaires with minimal assistance required from a family member.

Exclusion Criteria:

* Patients with head and neck cancer who have a treatment plan only including single modality therapy (ie just radiation, just surgery, or just systemic therapy)
* Patients who cannot speak, read and write in English with minimal assistance from a family member.
* Patients with cognitive impairment that would preclude the patient signing informed consent or understanding the materials.
* Patients who will not be receiving their cancer treatment at MGH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Information Satisfaction Questionnaire (ISQ) | Baseline, 4 Months, 6 Months
  The primary endpoint will be the difference in scores on the Information Satisfaction Questionnaire (ISQ) between participants in Phase I and Phase II at 3 weeks into their treatment.

SECONDARY OUTCOMES:
Percentage of participant change of scores of psychological distress | Baseline, 4 Months, 6 Months
Percentage of change participant symptom burden | Baseline, 4 Months, 6 Months
Percentage of Participant illness perception | Baseline, 4 Months, 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wirth, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States